CLINICAL TRIAL: NCT01419457
Title: A Phase I, Open-Label, Parallel-Group, Multiple-Dose Study to Determine the Pharmacokinetics of Favipiravir in Volunteers With Hepatic Impairment and in Healthy Control Volunteers
Brief Title: Pharmacokinetics of Favipiravir in Volunteers With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MDVI, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: T705aUS109
Record Dates: First submitted 2011-08-10; First posted 2011-08-18 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Healthy; Hepatic Impairment
Keywords: Healthy; hepatic impairment; T-705a; Favipiravir
MeSH Terms: interventions — favipiravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Experimental): Normal hepatic function
  Interventions: Drug: Favipiravir
- Group 2 (Experimental): Mild hepatic impairment
  Interventions: Drug: Favipiravir
- Group 3 (Experimental): Moderate hepatic impairment
  Interventions: Drug: Favipiravir
- Group 4 (Experimental): Severe hepatic impairment
  Interventions: Drug: Favipiravir

INTERVENTIONS:
Drug: Favipiravir — 1200 mg BID for Day 1 + 800 mg BID for Day 2-5
  Other Names: T-705a
  Arms: Group 1; Group 2; Group 3
Drug: Favipiravir — 800 mg BID for Day 1 + 400 mg BID for Day 2-3
  Other Names: T-705a
  Arms: Group 1; Group 4
Drug: Favipiravir — 800 mg Single Dose
  Arms: Group 4

SUMMARY:
This study is designed to determine the pharmacokinetics of favipiravir in volunteers with hepatic impairment and in healthy control volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Hepatically impaired groups:

  * Agree to doctor approved birth control methods from Day 1 until 3 months following the final dose of study drug.
  * Have mild hepatic impairment (Child-Pugh Clinical Assessment Score Grade A, score 5 6) or moderate hepatic impairment (Child-Pugh Clinical Assessment Score Grade B, score 7-9) or severe hepatic impairment (Child-Pugh Clinical Assessment Score Grade C, score 10-15);
* Control group

  * Agree to doctor approved birth control methods from Day 1 until 3 months following the final dose of study drug.
  * Healthy as determined by medical history, physical exam, vital signs, ECGs, and clinical laboratory tests.

Exclusion Criteria:

* Hepatically impaired groups:

  * Have used any drugs known to significantly affect hepatic metabolism within 28 days, or is unable or unwilling to forgo the use of such products throughout the study;
  * Have any acute or unstable condition or disease, other than impaired hepatic function, as determined by medical history, physical exam, ECG and clinical laboratory tests;
  * Known ongoing alcohol and/or drug abuse within 1 month
  * Any evidence of progressive worsening liver function disease as indicated by laboratory values;
  * Have had an acute flare of hepatitis A or B within 6 months;
  * Have acute, fulminant alcoholic hepatitis, determined either clinically or by histology;
  * Have a history of hepatoma or metastatic disease of the liver;
* Control group:

  * Have used any drugs known to significantly affect hepatic metabolism within 28 days, or is unable or unwilling to forgo the use of such products throughout the study;
  * Have a history or presence of clinically cardiovascular, dermatologic, endocrine, gastrointestinal, hematologic, hepatic, immunologic, neurologic, oncologic, psychiatric, pulmonary, or renal disease or any other condition.

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-08; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Cmax of favipiravir | predose and 0.25, 0.5, 0.75, 1, 2, 4, 6, 12, 18, 24, 36, 48 hours post-dose on Day 1 and Day 5
  The PK parameters for favipiravir and its metabolite in hepatically impaired adult subjects relative to healthy adult subjects matched for age, weight, gender, and race status on Day 1 and on Day 5.
AUC of favipiravir | predose and 0.25, 0.5, 0.75, 1, 2, 4, 6, 12, 18, 24, 36, 48 hours post-dose on Day 1 and Day 5
  The PK parameters for favipiravir and its metabolite in hepatically impaired adult subjects relative to healthy adult subjects matched for age, weight, gender, and race status on Day 1 and on Day 5.

SECONDARY OUTCOMES:
vital signs | 13 days
electrocardiograms [ECGs] | 13 days
clinical laboratory assessment | 13 days
adverse events [AEs] | 13 days
physical examination | 13 days

CONTACTS AND LOCATIONS:
Overall Officials: Richard A. Preston, MD/MSHP/MBA, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - University of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida